CLINICAL TRIAL: NCT03656874
Title: A Clinic-randomized Trial of a Clinical Decision Support System to Improve Dental Provider Delivery of Brief Tobacco Interventions and Quitline Referrals
Brief Title: Engaging Patients in Tobacco Cessation Resources in Dental Settings
Acronym: ENGAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); University of Sydney (Other); University of Pittsburgh (Other); Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: A15-107; U01DE026135 (NIH)
Record Dates: First submitted 2018-08-31; First posted 2018-09-04 (Actual); Results first posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-03

CONDITIONS: Smoking
Keywords: Decision Support Systems, Clinical; Smoking reduction; Smoking cessation; Smoking, Tobacco
MeSH Terms: conditions — Smoking; Smoking Reduction; Smoking Cessation; Tobacco Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Usual care, practitioners review clinical guidelines for tobacco during consent process.
- Clinical Decision Support (Experimental): The clinical decision support will provide clinical practice guideline-supported, evidence-based, and personalized scripts that are tailored based on patients' self-reported smoking attributes to deliver interventions consistent with the standard of care.
  Interventions: Other: Clinical Decision Support

INTERVENTIONS:
Other: Clinical Decision Support — The clinical decision support will provide clinical practice guideline-supported, evidence-based, and personalized scripts that are tailored based on patients' self-reported smoking attributes to deliver interventions consistent with the standard of care
  Arms: Clinical Decision Support

SUMMARY:
The overarching goal of this project is to reduce smoking-associated morbidity and mortality by increasing the number of patients who are referred for tobacco cessation counseling. Using a stratified, group-randomized, controlled, 2-arm trial conducted in two settings, the investigators will compare smoking-related clinical decision support (CDS) to usual care.

DETAILED DESCRIPTION:
This project aims to reduce smoking-associated morbidity and mortality by increasing the number of patients who are referred for tobacco cessation counseling. The study team will evaluate the effectiveness of clinical decision support (CDS) to improve dental provider delivery of brief tobacco interventions and referrals to tobacco quitlines for further tobacco counseling. The CDS will generate personalized, evidence-based recommendations for dentists and dental hygienists to actively engage their smoking patients in the course of usual dental care. Subsequently, the study team will assess the tobacco cessation actions of smokers using patient-centered outcomes.

ELIGIBILITY:
DENTAL STUDENTS AND DENTAL HYGIENE STUDENTS

Inclusion Criteria:

* 3rd and 4th year predoctoral students or dental hygiene students enrolled at selected dental schools

PRIVATE PRACTICE DENTISTS & HYGIENISTS

Inclusion Criteria:

* General practice dentists or dental hygienists practicing at selected private practice clinics

Exclusion Criteria:

* Providers not able or willing to record current tobacco use status in their electronic health record
* Providers affiliated with selected dental schools who hold a current teaching or clinical position

PATIENTS

Inclusion Criteria:

* Current cigarette smokers

Exclusion Criteria:

* patients requesting to opt out of research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: D. Brad Rindal, DDS, Principal Investigator — HealthPartners Institute; Heiko Spallek, DMD,PhD,MSBA, Principal Investigator — University of Sydney
Locations (3):
- United States (3):
  - Indiana University School of Dentistry, Indianapolis, Indiana
  - HealthPartners Institute, Bloomington, Minnesota
  - University of Pittsburgh School of Dental Medicine, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Sharing of study outputs and resources is an essential element of this research. To facilitate the conduct of future research, we will make available de-identified datasets and technical resources from the completed project in a manner consistent with human subject protection and HIPAA privacy regulations. These resources will be subject to requirements imposed by the governing Institutional Review Board (IRB) and our organizational legal requirements.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Release of de-identified datasets and accompanying technical resources used for specific publications will occur within 6 months of the online publication date.
Access Criteria: Data will be stored at HealthPartners Institute by the project co-principal investigator/site lead and statistician. Study publications will note the method for requesting the study data and technical materials. The study statistician will provide data and accompanying files in an archived zip format to requesters via email. Data will not be stored in a public repository.

REFERENCES:
- [Derived] Holliday R, Hong B, McColl E, Livingstone-Banks J, Preshaw PM. Interventions for tobacco cessation delivered by dental professionals. Cochrane Database Syst Rev. 2021 Feb 19;2(2):CD005084. doi: 10.1002/14651858.CD005084.pub4. PMID 33605440

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study took place at two academic institutions and private practices in the community. Due to technical difficulties regarding the implementation of the Clinical Decision Support (CDS) tool into the school's electronic dental record, the two academic institutions were discontinued from the study. Private practice clinics in the community were the focus of the ongoing study with clinic randomization occurring between March 29, 2019 and December 30, 2019 for 9 months.
Pre-assignment Details: Randomization occurred at the clinic level.107 patients were authorized at their dental clinic to be contacted for the study. 51 patients declined to be consented or were not able to be reached; 56 participants consented to participate in the study.
Units Other Than Participants: Clinics
Groups:
- Clinical Decision Support: Clinical decision support will provide clinical practice guideline-supported, evidence-based, and personalized scripts that are tailored based on patients' self-reported smoking attributes to deliver interventions consistent with the standard of care.
Period: Overall Study
Arm/Group | Usual Care | Clinical Decision Support
Started (Patient Participants) | 13; 4 Clinics | 43; 6 Clinics
Completed (Patient participants) | 10; 2 Clinics | 26; 5 Clinics
Not Completed | 3; 2 Clinics | 17; 1 Clinics
Not completed — Lost to Follow-up | 3 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Clinical Decision Support | Total
Number analyzed (Participants) | 13 | 43 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 43 | 56
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (19.2) | 41.8 (14.9) | 42.3 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 35 | 40
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 13 | 40 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 9 | 9
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 11 | 31 | 42
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 43 | 56

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Smokers With Delivery of Brief Interventions and/or Referral to Treatment
Description: Composite of provider actions reported by patient regarding delivery of brief interventions and/or referral to treatment. These actions included that the provider 1) delivered a brief smoking intervention by discussing, a)developing a quit plan or b)setting a quit date or c)using medications to help patients quit or d)discussed strategies for quitting. The provider made a 2) referral to a quitline; a)provided information about how to contact a tobacco quitline or b) arranged for the patient to be contacted by the tobacco quit line for smoking cessation. The composite is satisfied if the patient reports that any of the intervention activities or referral was delivered by the provider.
Time Frame: within a week of the index dental encounter
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Clinical Decision Support
Number analyzed (Participants) | 13 | 43
Participants | 7 | 36

2. Secondary Outcome: Percentage of Smokers With Initial Actions Related to Cessation
Description: Composite of patient-reported actions of smokers with initial actions related to cessation. This composite is met if the patient reported that they contacted a smoking cessation quitline, set a quit date, developed a plan to quit, or is starting nicotine replacement or other medication to help quit within 1-7 days of their index dental visit.
Time Frame: within a week of index dental encounter
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Clinical Decision Support
Number analyzed (Participants) | 13 | 43
Participants | 3 | 20

3. Secondary Outcome: Percentage of Smokers With Long-term Actions Related to Cessation
Description: Composite of patient-reported actions of smokers with long-term actions related to cessation. This composite includes whether the patient reported that they quit smoking (stopped smoking for more than one day because they were trying to stop smoking), or reduced their smoking use (50% reduction in amount smoked at 6 months compared to baseline). This composite is satisfied if the patient reports that they have done any of these actions within the 6 months +/- 1 week period between the index dental visit and the date of the second patient survey.
Time Frame: within six-months of index dental encounter
Population: The numbers represented here indicate that not all study participants completed questionnaires at 6 months and were lost to follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Clinical Decision Support
Number analyzed (Participants) | 10 | 26
Participants | 4 | 18

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Usual Care | Clinical Decision Support
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/43
Other Adverse Events (participants affected / at risk) | 0/13 | 0/43

LIMITATIONS AND CAVEATS:
Technological interface issues and coronavirus disease (COVID) were limitations of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-01-12): https://cdn.clinicaltrials.gov/large-docs/74/NCT03656874/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/74/NCT03656874/SAP_001.pdf
  • Informed Consent Form (2019-11-21): https://cdn.clinicaltrials.gov/large-docs/74/NCT03656874/ICF_002.pdf